CLINICAL TRIAL: NCT00453388
Title: Nonmyeloablative Hematopoietic Cell Transplantation for Patients With Fanconi Anemia Using Alternative Marrow Donors: A Phase II Dose-Finding Study
Brief Title: Fludarabine Phosphate, Cyclophosphamide, and Total-Body Irradiation Followed by Donor Bone Marrow Transplant, Mycophenolate Mofetil, and Cyclosporine in Treating Patients With Fanconi Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2064.00; NCI-2010-00238 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2064.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2019-12

CONDITIONS: Acute Myeloid Leukemia in Remission; de Novo Myelodysplastic Syndrome; Fanconi Anemia; Previously Treated Myelodysplastic Syndrome
MeSH Terms: conditions — Fanconi Anemia | interventions — Cyclophosphamide; Cyclosporine; Cyclosporins; fludarabine phosphate; Mycophenolic Acid; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (2 vs 2.5 vs 3 Gy TBI dose-escalation) (Experimental): Patients with a history of hematologic malignancy and HLA-haploidentical donor receive fludarabine phosphate (FLU) intravenously (IV) over 1 hour on days -6 to -2, and undergo TBI on day -1 and allogeneic bone marrow transplant on day 0. Patients then receive CY IV over 1 hour on days 3 and 4, MMF orally (PO) thrice daily (TID) on days 5-35, and CSP IV or PO on days 5-84, with taper until day 180, in the absence of GVHD.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Drug: Cyclophosphamide; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Radiation: Total-Body Irradiation
- Arm II (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI de-escalation) (Experimental): Patients with no history of hematological malignancy and HLA-haploidentical donors receive FLU IV over 1 hour on days -6 to -2, and undergo TBI on day -1 and allogeneic bone marrow transplant on day 0. Patients then receive CY IV over 1 hour on days 3 and 4, MMF PO TID on days 5-35, and CSP IV or PO on days 5-84, with taper until day 180, in the absence of GVHD.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Drug: Cyclophosphamide; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Radiation: Total-Body Irradiation
- Arm III (2 vs 2.5 vs 3 Gy TBI dose-escalation) (Experimental): Patients with history of hematologic malignancy and HLA-matched unrelated donors receive FLU IV over 1 hour on days -6 to -2, and undergo TBI on day -1 and allogeneic bone marrow transplant on day 0. Patients then receive CY IV over 1 hour on days 3 and 4, MMF PO TID on days 5-35, and CSP IV or PO on days 5-84, with taper until day 180, in the absence of GVHD.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Drug: Cyclophosphamide; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Radiation: Total-Body Irradiation
- Arm IV (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI de-escalation) (Experimental): Patients with no history of hematological malignancy and HLA-matched unrelated donors receive FLU IV over 1 hour on days -6 to -2, and undergo TBI on day -1 and allogeneic bone marrow transplant on day 0. Patients then receive CY IV over 1 hour on days 3 and 4, MMF PO TID on days 5-35, and CSP IV or PO on days 5-84, with taper until day 180, in the absence of GVHD.
  Interventions: Procedure: Allogeneic Bone Marrow Transplantation; Drug: Cyclophosphamide; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Bone Marrow Transplantation — Undergo allogeneic bone marrow transplant
  Other Names: Allo BMT; Allogeneic BMT
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cyclosporine — Given IV or PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; Oforta; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic stem cell transplant
  Other Names: Non-myeloablative allogeneic transplant; Nonmyeloablative Stem Cell Transplantation; NST
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This phase II trial studies how well total-body irradiation (TBI) works when given together with fludarabine phosphate and cyclophosphamide followed by donor bone marrow transplant, mycophenolate mofetil, and cyclosporine in treating patients with Fanconi anemia (FA). Giving low doses of chemotherapy, such as fludarabine phosphate and cyclophosphamide, and TBI before or after a donor bone marrow transplant helps stop the growth of abnormal cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving mycophenolate mofetil and cyclosporine after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify doses of total-body irradiation (TBI) that lead to sufficient probability of donor engraftment (> 5% donor cluster of differentiation [CD]3 chimerism) by day +200.

II. Evaluate the probability of severe acute graft-versus-host disease.

SECONDARY OBJECTIVES:

I. Evaluate the probabilities of overall survival, regimen-related toxicity (RRT), and recurrent hematopoietic malignancy in those patients with a prior underlying history of such.

II. Examine the degree to which mixed chimerism provides for amelioration of symptoms (i.e., infections due to neutropenia, hemorrhage due to thrombocytopenia) associated with bone marrow failure.

III. Determine if the FA complementation group and % initial mosaicism predict engraftment and RRT outcomes.

OUTLINE: Patients are assigned to 1 of 4 treatment arms.

NOTE: Patients no longer receive pre-transplant cyclophosphamide as of February 2009.

After completion of study treatment, patients are followed up at 6 months and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with FA and bone marrow (BM) failure involving 2 of the following 3 lineages: granulocyte count < 0.5 x 10^9/L, platelet count < 20 x 10^9/L, or hemoglobin < 8 g/dL
* Any patient with FA who requires red blood cell or platelet transfusions because of marrow failure
* Any patient with FA who has a life-threatening BM failure involving a single hematopoietic lineage
* Any patient with FA and pre-existing cytogenetic abnormality including hematopoietic malignancy (acute myeloid leukemia [AML] or myelodysplastic syndrome [MDS]) in morphological remission (defined as absence of circulating blasts and bone marrow blasts < 5% as assessed by morphology); Note that hematopoietic recovery is not required for remission status
* Patients must have a negative cytotoxic cross match with donor
* DONOR: Related, human leukocyte antigen (HLA)-haploidentical donors must be identical for one HLA haplotype and mismatched for any number of HLA-A, -B, -C, DRB1 or DQB1 loci of the unshared haplotype
* DONOR: Unrelated, HLA-matched donors must be matched at HLA-A, B, C, DRB1 and DQB1 by deoxyribonucleic acid (DNA) typing at the highest resolution routinely available at the time of donor selection; a single allele mismatch at HLA-A, B, or C is allowed OR a single DQB1 mismatch is allowed
* DONOR: Bone marrow will be the only allowed hematopoietic stem cell source
* DONOR: Haploidentical donor selection will be based on standard institutional criteria, otherwise no specific prioritization will be made amongst the suitable available donors

Exclusion Criteria:

* Patients having available HLA-matched related donors
* Significant organ dysfunction that would prevent compliance with conditioning, graft-versus-host disease (GVHD) prophylaxis, or would severely limit the probability of survival, such as liver disease/failure (active hepatitis, moderate to severe portal fibrosis/cirrhosis confirmed by biopsy or uncorrectable hepatic synthetic dysfunction), lung disease, or cardiac disease (ejection fraction < 35%, or if unable to obtain ejection fraction, shortening fraction of < 26%; if shortening is < 26% a cardiology consult is required with principal investigator [PI] having final approval of eligibility)
* Human immunodeficiency virus (HIV) seropositive patients
* Fertile females who are unwilling to use contraceptive techniques during and for the twelve months following treatment, as well as females who are pregnant or actively breast feeding
* Fertile males who are unwilling to use contraceptive techniques during and for the twelve months following treatment
* AML/MDS in morphological relapse, defined as having circulating blasts or bone marrow blasts >= 5% as assessed by morphology
* Active infectious disease concerns
* Karnofsky performance score < 50 or Lansky performance score < 40
* DONOR: Donors found to have Fanconi anemia based on chromosomal breakage analysis
* DONOR: Donors who are not expected to meet the minimum target dose of marrow cells (1 x 10^8 nucleated cells/kg recipient ideal body weight [IBW]) or who are unwilling to be bone marrow donors
* DONOR: HIV-positive donors
* DONOR: Donors who are cross-match positive with recipient
* DONOR: Recipient homozygous at mismatched locus; if the recipient is homozygous at HLA-A, B, or C and the donor is mismatched at that locus, the donor should be avoided; exceptions must be discussed with the PI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Kiem, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (5):
- United States (4):
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Universidade Federal do Paraná, Curitiba, Paraná, Brazil

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (2 vs 2.5 vs 3 Gy TBI Dose-escalation) | Arm II (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation) | Arm III (2 vs 2.5 vs 3 Gy TBI Dose-escalation) | Arm IV (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation)
Started | 0 | 5 | 1 | 0
Completed | 0 | 5 | 1 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects meeting the criteria for Arms I or IV were enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (2 vs 2.5 vs 3 Gy TBI Dose-escalation) | Arm II (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation) | Arm III (2 vs 2.5 vs 3 Gy TBI Dose-escalation) | Arm IV (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation) | Total
Number analyzed (Participants) | 0 | 5 | 1 | 0 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 5 | 1 |  | 6
  Between 18 and 65 years |  | 0 | 0 |  | 0
  >=65 years |  | 0 | 0 |  | 0
Age, Continuous [Median (Full Range); unit: years] |  | 11.1 [6.9 to 13.9] | 11.9 [11.9 to 11.9] |  | 11.1 [6.9 to 13.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 5 | 0 |  | 5
  Male |  | 0 | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 3 | 1 |  | 4
  Brazil |  | 2 | 0 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Engraft at Each Dose of TBI Used
Description: Number of subjects who engrafted. Engraftment defined as greater than 95% donor chimerism.
Time Frame: Up to Day 200
Population: No subjects meeting the criteria for Arms I or IV were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (2 vs 2.5 vs 3 Gy TBI Dose-escalation) | Arm II (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation) | Arm III (2 vs 2.5 vs 3 Gy TBI Dose-escalation) | Arm IV (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation)
Number analyzed (Participants) | 0 | 5 | 1 | 0
Participants |  | 5 | 1 |

2. Primary Outcome: Incidence of Grades III-IV Acute GVHD
Description: Number of subjects who developed maximum grade acute graft-vs-host disease
  aGVHD Stages
  Skin:
  1. - a maculopapular eruption involving < 25% BSA
  2. - a maculopapular eruption involving 25 - 50% BSA
  3. - generalized erythroderma
  4. - generalized erythroderma with bullous formation and often with desquamation
  Liver:
  1. - bilirubin 2.0 - 3.0 mg/100 mL
  2. - bilirubin 3 - 5.9 mg/100 mL
  3. - bilirubin 6 - 14.9 mg/100 mL
  4. - bilirubin > 15 mg/100 mL
  Gut:
  Diarrhea is graded 1 - 4 in severity. Nausea and vomiting and/or anorexia caused by GVHD is assigned as 1 in severity. The severity of gut involvement is assigned to the most severe involvement noted. Patients with visible bloody diarrhea are at least stage 2 gut and grade 3 overall.
  aGVHD Grades Grade III: Stage 2 - 4 gastrointestinal involvement and/or +2 to +4 liver involvement, with or without a rash Grade IV: Pattern and severity of GVHD similar to grade 3 with extreme constitutional symptoms or death
Time Frame: Up to Day 100
Population: No subjects meeting the criteria for Arms I or IV were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (2 vs 2.5 vs 3 Gy TBI Dose-escalation) | Arm II (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation) | Arm III (2 vs 2.5 vs 3 Gy TBI Dose-escalation) | Arm IV (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation)
Number analyzed (Participants) | 0 | 5 | 1 | 0
Participants |  | 1 | 0 |

3. Secondary Outcome: Incidence of Transplant-related Mortality
Description: Number of subjects who expired due to transplant-related mortality
Time Frame: Up to Day 200
Population: No subjects meeting the criteria for Arms I or IV were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (2 vs 2.5 vs 3 Gy TBI Dose-escalation) | Arm II (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation) | Arm III (2 vs 2.5 vs 3 Gy TBI Dose-escalation) | Arm IV (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation)
Number analyzed (Participants) | 0 | 5 | 1 | 0
Participants |  | 1 | 0 |

4. Secondary Outcome: Incidence of Adverse Events
Description: Number of subjects who developed reportable AEs, assessed using adapted version of the Common Toxicity Criteria
Time Frame: Up to Day 100
Population: No subjects meeting the criteria for Arms I or IV were enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (2 vs 2.5 vs 3 Gy TBI Dose-escalation) | Arm II (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation) | Arm III (2 vs 2.5 vs 3 Gy TBI Dose-escalation) | Arm IV (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation)
Number analyzed (Participants) | 0 | 5 | 1 | 0
Participants |  | 3 | 0 |

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200
Description: No subjects meeting the criteria for Arms I or IV were enrolled.
Arm/Group | Arm I (2 vs 2.5 vs 3 Gy TBI Dose-escalation) | Arm II (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation) | Arm III (2 vs 2.5 vs 3 Gy TBI Dose-escalation) | Arm IV (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation)
All-Cause Mortality (participants affected / at risk) | 0/0 | 2/5 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 2/5 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 3/5 | 0/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (2 vs 2.5 vs 3 Gy TBI Dose-escalation) (N=0) | Arm II (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation) (N=5) | Arm III (2 vs 2.5 vs 3 Gy TBI Dose-escalation) (N=1) | Arm IV (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation) (N=0)
Death (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Septic shock
severe abdominal pain associated with GVHD (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (2 vs 2.5 vs 3 Gy TBI Dose-escalation) (N=0) | Arm II (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation) (N=5) | Arm III (2 vs 2.5 vs 3 Gy TBI Dose-escalation) (N=1) | Arm IV (2 vs 2.5 vs 3 vs 1 vs 0 Gy TBI De-escalation) (N=0)
Mucositis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0
elevated bilitrubin (Hepatobiliary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
pulmonary hemorrage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes